CLINICAL TRIAL: NCT00892723
Title: A Pilot Phase 2a Blinded, Placebo Controlled, Multicenter Parallel Group, Dose Ranging Study to Evaluate the Safety and Preliminary Efficacy of Additional Doses of AZX100 Drug Product Following Excision of Keloids
Brief Title: A Study to Evaluate the Safety and Efficacy of Additional Doses of AZX100 Drug Product Following Excision of Keloid Scars
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capstone Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OL-ASCAR-05
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-09

CONDITIONS: Scar Prevention; Scar Reduction
Keywords: AZX100; Patient and Observer Scar Assessment Scale; POSAS; Visual Analog Scale; VAS; Keloid; Scarring; Scar reduction; Scar prevention
MeSH Terms: conditions — Keloid; Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Experimental)
  Interventions: Drug: AZX100 Drug Product
- High Dose (Experimental)
  Interventions: Drug: AZX100 Drug Product
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZX100 Drug Product — Subjects were administered AZX100 0.3 mg per linear centimeter (low dose) intradermally at the site of the keloid scar removal. The first dose was given 19-23 days following surgery, and the second dose was given 40-44 days following surgery.
  Arms: Low Dose
Drug: Placebo — Subjects were administered placebo (0.9% saline) per linear centimeter intradermally at the site of the keloid scar removal. The first dose was given 19-23 days following surgery, and the second dose was given 40-44 days following surgery.
  Arms: Placebo
Drug: AZX100 Drug Product — Subjects were administered AZX100 10 mg per linear centimeter (high dose) intradermally at the site of the keloid scar removal. The first dose was given 19-23 days following surgery, and the second dose was given 40-44 days following surgery.
  Arms: High Dose

SUMMARY:
The purpose of this study was to determine the safety of AZX100 Drug Product and to determine whether it was effective in preventing or reducing re-growth of surgically removed keloid scars.

ELIGIBILITY:
Inclusion Criteria:

* Keloid scar located below the neck between 1 and 3 cm long and less than 1 cm at its widest point
* Willing to undergo keloid scar excision surgery
* Healthy adult male or non-pregnant female
* Non-diabetic
* Body Mass Index in the range of 18-35
* No clinically significant abnormal values on a full blood safety screen
* Non-smoker and non-nicotine user for the previous six months

Exclusion Criteria:

* History or clinical evidence of acute or chronic disease
* History of cancer within the last 5 years, except for surgically removed cancers of the skin that are not near the keloid area
* History of anaphylactic shock or anaphylactoid (hypersensitivity) reaction
* Allergy to local anesthesia, including lidocaine and epinephrine
* Dermatologic disorders, except for folliculitis and acne
* On therapy with steroids
* On therapy with a drug that would affect collagen synthesis
* Positive urine test for nicotine or drugs of abuse
* Positive blood test for HIV 1 or 2, hepatitis B or hepatitis C
* Positive blood test for anti-AZX100 antibodies
* Participation in another study within 60 days prior to enrollment
* Blood donation within 7 days before dosing with study drug
* Plasma donation within 3 days before dosing with study drug
* Tattoo within approximately 3 cm of the keloid scar that will be removed
* Apply any lotion or cream on or near the keloid scar that will be removed within 14 days before dosing with study drug
* Use of a tanning bed or tanning light within the 3 months before enrollment
* Intend to use any scar improving product during of the study (1 year)
* History of drug addiction or excessive use of alcohol
* Previous drug treatment of the keloid scar within the last 3 years, or have had any laser, irradiation, or surgical treatment of the keloid scar that will be removed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lotus Clinical Research, Inc., Pasadena, California
  - Paddington Testing Company, Inc., Philadelphia, Pennsylvania
  - DermResearch, Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the study began in June 2009 and was completed in September 2010. All patients were enrolled in dermatological medical clinics.
Groups:
- Low Dose: AZX100 Drug Product 0.3 mg was administered intradermally per linear centimeter along the excision line following keloid scar excision at 21 days and 42 days after surgery.
- High Dose: AZX100 Drug Product 1 mg was administered intradermally per linear centimeter along the excision line following keloid scar excision at 21 days and 42 days after surgery.
- Placebo: Placebo (0.9% saline) was administered intradermally per linear centimeter along the excision line following keloid scar excision at 21 days and 42 days after surgery.
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 21 | 19 | 19
Completed | 19 | 15 | 17
Not Completed | 2 | 4 | 2
Not completed — Lost to Follow-up | 1 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 21 | 19 | 19 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 19 | 59
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.1 (11) | 36.1 (10.9) | 37.5 (12.4) | 36.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 7 | 25
  Male | 10 | 12 | 12 | 34
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Differences Among the 3 Dosage Groups in the Patient (PSAS) and Observer (OSAS) Scar Assessment Scale (POSAS) Scores
Description: Efficacy was based on the difference between mean POSAS scores of placebo, 0.3 mg AZX100, and 1 mg AZX100 12 months after surgery. This gave four comparisons to placebo: patient or observer and 0.3 mg and 1 mg AZX100. PSAS included patients' ratings on a scale of 1-10 (1 was normal skin or no complaints and 10 was the worst imaginable scar or the worst difference) for the following: Is the scar painful? Is the scar itching? Is the color of the scar different? Is the scar more stiff? Is the thickness of the scar different? Is the scar irregular? The possible minimum score was 6 and the maximum (worst) score was 60. OSAS included observers' ratings on a scale of 1-10 (1 was normal skin and 10 was the worst scar imaginable) for vascularization, pigmentation, thickness, relief, and pliability. The possible minimum score was 5 and the possible maximum (worst) score was 50.
Time Frame: 12 Months
Population: In this early phase study, the efficacy and safety analyses were performed using an evaluable subject sample, which included all subjects who received study agent and provided some efficacy or safety data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PSAS Results for Placebo: This group included Month 12 PSAS scores for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- PSAS Results for 0.3 mg AZX100: This group included Month 12 PSAS scores for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- PSAS Results for 1 mg AZX100: This group included Month 12 PSAS scores for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- OSAS Results for Placebo: This group included Month 12 OSAS scores for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- OSAS Results for 0.3 mg AZX100: This group included Month 12 OSAS scores for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- OSAS Results for 1 mg AZX100: This group included Month 12 OSAS scores for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
Arm/Group | PSAS Results for Placebo | PSAS Results for 0.3 mg AZX100 | PSAS Results for 1 mg AZX100 | OSAS Results for Placebo | OSAS Results for 0.3 mg AZX100 | OSAS Results for 1 mg AZX100
Number analyzed (Participants) | 19 | 21 | 19 | 19 | 21 | 19
Units on a scale | 23.29 (15.06) | 24.11 (14.75) | 21.33 (11.36) | 18.53 (10.07) | 23.47 (8.78) | 18.33 (10.00)
Statistical Analysis 1: Comparison: PSAS Results for Placebo vs PSAS Results for 0.3 mg AZX100; Test type: Superiority or Other; p = 0.87, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 2: Comparison: PSAS Results for Placebo vs PSAS Results for 1 mg AZX100; Test type: Superiority or Other; p = 0.86, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 3: Comparison: OSAS Results for Placebo vs OSAS Results for 0.3 mg AZX100; Test type: Superiority or Other; p = 0.11, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 4: Comparison: OSAS Results for Placebo vs OSAS Results for 1 mg AZX100; Test type: Superiority or Other; p = 0.91, Wilcoxon (rank sum); For this early phase study, no adjustment was used

2. Secondary Outcome: Between-group Mean Differences in Visual Analog Scale (VAS) Scores by Independent Blinded Raters
Description: At 12 months, two independent dermatologists who were blinded to study treatment evaluated the scar images using a Visual Analog Scale (VAS) of 0-100 mm, with 0 being normal skin and 100 being the worst scar imaginable. The scars were presented in a scrambled order. Efficacy was based on the difference between VAS scores of placebo and 0.3 mg AZX100, and placebo and 1 mg AZX100, for each of the two raters separately. Data from the two raters was not combined.
Time Frame: 12 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters
Groups:
- Rater 1 VAS Scores for Placebo; Rater 2 VAS Scores for Placebo: This group included Month 12 VAS scores for those patients who received placebo (saline)/linear centimeter intradermally along the excision line following keloid scar excision at 21 days and 42 days after surgery.
- Rater 1 VAS Scores for 0.3 mg AZX100; Rater 2 VAS Scores for 0.3 mg AZX100: This group included Month 12 VAS scores for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line following keloid scar excision at 21 days and 42 days after surgery.
- Rater 1 VAS Scores for 1 mg AZX100; Rater 2 VAS Scores for 1 mg AZX100: This group included Month 12 VAS scores for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line following keloid scar excision at 21 days and 42 days after surgery.
Arm/Group | Rater 1 VAS Scores for Placebo | Rater 1 VAS Scores for 0.3 mg AZX100 | Rater 1 VAS Scores for 1 mg AZX100 | Rater 2 VAS Scores for Placebo | Rater 2 VAS Scores for 0.3 mg AZX100 | Rater 2 VAS Scores for 1 mg AZX100
Number analyzed (Participants) | 19 | 21 | 19 | 19 | 21 | 19
Millimeters | 71.9 (21.2) | 77.0 (20.3) | 68.1 (23.3) | 56.1 (12.8) | 62.2 (10.9) | 54.3 (13.2)
Statistical Analysis 1: Comparison: Rater 1 VAS Scores for Placebo vs Rater 1 VAS Scores for 0.3 mg AZX100; Test type: Superiority or Other; p = 0.23, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 2: Comparison: Rater 1 VAS Scores for Placebo vs Rater 1 VAS Scores for 1 mg AZX100; Test type: Superiority or Other; p = 0.82, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 3: Comparison: Rater 2 VAS Scores for Placebo vs Rater 2 VAS Scores for 0.3 mg AZX100; Test type: Superiority or Other; p = 0.23, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 4: Comparison: Rater 2 VAS Scores for Placebo vs Rater 2 VAS Scores for 1 mg AZX100; Test type: Superiority or Other; p = 0.71, Wilcoxon (rank sum); For this early phase study, no adjustment was used

3. Secondary Outcome: Between-group Mean Differences in Objective Measures Obtained Via 3D Photography (Elevation, Length, Width)
Description: This secondary outcome included measurements based on 3D photography of the scar surface at Month 12 and included maximum length, maximum width perpendicular to the maximum length, and minimum, maximum and mean elevation. All elevation measurements were made relative to the interpolated smooth skin surface. A value closest to zero was preferred, because zero was equal to the normal skin surface. The minimum elevation value was calculated as the lowest point of the scar below the interpolated smoooth skin surface and was always a negative number. A more negative number was worse, because it indicated a deeper measurement below the interpolated smooth skin surface. The maximum elevation value was calculated as the highest point of the scar above the interpolated smooth skin surface. A larger number was worse because it indicated a higher peak above the interpolated smooth skin surface. The mean elevation of the scar relative to the interpolated smooth skin surface was also calculated.
Time Frame: 12 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters
Groups:
- Scar Length - Placebo: This group included Month 12 scar length measurements (mm)for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Length - 0.3 mg AZX100: This group included Month 12 scar length measurements (mm) for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Length - 1 mg AZX100: This group included Month 12 scar length measurements (mm) for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Width - Placebo: This group included Month 12 scar width measurements (mm) for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Width - 0.3 mg AZX100: This group included Month 12 scar width measurements (mm) for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Width - 1 mg AZX100: This group included Month 12 scar width measurements (mm)for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Minimum Elevation - Placebo: This group included Month 12 scar minimum elevation measurements (mm) for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Minimum Elevation - 0.3 mg AZX100: This group included Month 12 scar minimum elevation measurements (mm) for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Minimum Elevation - 1 mg AZX100: This group included Month 12 scar minimum elevation measurements f(mm) or those patients who received 1 mg/ AZX100linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Maximum Elevation - Placebo: This group included Month 12 scar maximum elevation measurements f(mm) or those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Maximum Elevation - 0.3 mg AZX100: This group included Month 12 scar maximum elevation measurements (mm) for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Maximum Elevation - 1 mg AZX100: This group included Month 12 scar maximum elevation measurements (mm) for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Mean Elevation - Placebo: This group included Month 12 scar mean elevation measurements (mm) for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Mean Elevation - 0.3 mg AZX100: This group included Month 12 scar mean elevation measurements (mm) for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Mean Elevation - 1 mg AZX100: This group included Month 12 scar mean elevation measurements (mm) for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
Arm/Group | Scar Length - Placebo | Scar Length - 0.3 mg AZX100 | Scar Length - 1 mg AZX100 | Scar Width - Placebo | Scar Width - 0.3 mg AZX100 | Scar Width - 1 mg AZX100 | Scar Minimum Elevation - Placebo | Scar Minimum Elevation - 0.3 mg AZX100 | Scar Minimum Elevation - 1 mg AZX100 | Scar Maximum Elevation - Placebo | Scar Maximum Elevation - 0.3 mg AZX100 | Scar Maximum Elevation - 1 mg AZX100 | Scar Mean Elevation - Placebo | Scar Mean Elevation - 0.3 mg AZX100 | Scar Mean Elevation - 1 mg AZX100
Number analyzed (Participants) | 19 | 21 | 19 | 19 | 21 | 19 | 19 | 21 | 19 | 19 | 21 | 19 | 19 | 21 | 19
Millimeters | 27.71 (6.76) | 27.90 (7.67) | 27.51 (5.63) | 13.48 (4.82) | 15.67 (5.03) | 12.52 (4.28) | -0.86 (1.09) | -0.57 (0.62) | -0.38 (0.12) | 2.01 (1.20) | 2.44 (1.36) | 1.74 (0.92) | 0.40 (0.40) | 0.51 (0.34) | 0.31 (0.25)
Statistical Analysis 1: Comparison: Scar Length - Placebo vs Scar Length - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.73, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 2: Comparison: Scar Length - Placebo vs Scar Length - 1 mg AZX100; Test type: Superiority or Other; p = 0.94, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 3: Comparison: Scar Width - Placebo vs Scar Width - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.14, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 4: Comparison: Scar Width - Placebo vs Scar Width - 1 mg AZX100; Test type: Superiority or Other; p = 0.68, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 5: Comparison: Scar Minimum Elevation - Placebo vs Scar Minimum Elevation - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.56, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 6: Comparison: Scar Minimum Elevation - Placebo vs Scar Minimum Elevation - 1 mg AZX100; Test type: Superiority or Other; p = 0.32, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 7: Comparison: Scar Maximum Elevation - Placebo vs Scar Maximum Elevation - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.33, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 8: Comparison: Scar Maximum Elevation - Placebo vs Scar Maximum Elevation - 1 mg AZX100; Test type: Superiority or Other; p = 0.65, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 9: Comparison: Scar Mean Elevation - Placebo vs Scar Mean Elevation - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.21, Wilcoxon (rank sum); For this early phase study, no adjustment was used
Statistical Analysis 10: Comparison: Scar Mean Elevation - Placebo vs Scar Mean Elevation - 1 mg AZX100; Test type: Superiority or Other; p = 0.90, Wilcoxon (rank sum); For this early phase study, no adjustment was used

4. Secondary Outcome: Between-group Mean Differences in Objective Measures Obtained Via 3D Photography (Volume)
Description: This secondary outcome included measurements based on 3D photography of the scar surface at Month 12 and included positive volume, negative volume and total volume. All volume measurements were made relative to the interpolated smooth skin surface. A value closer to zero was preferred, because zero was equal to the normal skin surface. Positive volume was calculated as the volume of the scar above the interpolated smooth skin surface. Negative volume was calculated as the volume of the scar below the interpolated smooth skin surface, and was always a negative number. Total volume was calculated as the sum of the positive volume and the absolute value of the negative volume.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters cubed
Groups:
- Scar Positive Volume - Placebo: This group included Month 12 scar positive volume measurements (mm^3) for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Positive Volume - 0.3 mg AZX100: This group included Month 12 scar positive volume measurements (mm^3) for those patients who received 0.3 mg AZx100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Positive Volume - 1 mg AZX100: This group included Month 12 scar positive volume measurements (mm^3) for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Negative Volume - Placebo: This group included Month 12 scar negative volume measurements (mm^3) for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Negative Volume - 0.3 mg AZX100: This group included Month 12 scar negative volume measurements (mm^3) for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Negative Volume - 1 mg AZX100: This group included Month 12 scar negative volume measurements (mm^3) for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Total Volume - Placebo: This group included Month 12 scar total volume measurements (mm^3) for those patients who received placebo (saline)/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Total Volume - 0.3 mg AZX100: This group included Month 12 scar total volume measurements (mm^3) for those patients who received 0.3 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
- Scar Total Volume - 1 mg AZX100: This group included Month 12 scar total volume measurements (mm^3) for those patients who received 1 mg AZX100/linear centimeter intradermally along the excision line at 21 days and 42 days after surgery.
Arm/Group | Scar Positive Volume - Placebo | Scar Positive Volume - 0.3 mg AZX100 | Scar Positive Volume - 1 mg AZX100 | Scar Negative Volume - Placebo | Scar Negative Volume - 0.3 mg AZX100 | Scar Negative Volume - 1 mg AZX100 | Scar Total Volume - Placebo | Scar Total Volume - 0.3 mg AZX100 | Scar Total Volume - 1 mg AZX100
Number analyzed (Participants) | 19 | 21 | 19 | 19 | 21 | 19 | 19 | 21 | 19
Millimeters cubed | 0.42 (0.39) | 0.65 (0.49) | 0.37 (0.25) | -0.04 (0.06) | -0.06 (0.07) | -0.06 (0.05) | 0.45 (0.39) | 0.71 (0.53) | 0.43 (0.23)
Statistical Analysis 1: Comparison: Scar Positive Volume - Placebo vs Scar Positive Volume - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.16, Wilcoxon (signed rank); For this early phase study, no adjustment was used
Statistical Analysis 2: Comparison: Scar Positive Volume - Placebo vs Scar Positive Volume - 1 mg AZX100; Test type: Superiority or Other; p = 0.74, Wilcoxon (signed rank) — For this early phase study, no adjustment was used
Statistical Analysis 3: Comparison: Scar Negative Volume - Placebo vs Scar Negative Volume - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.45, Wilcoxon (signed rank) — For this early phase study, no adjustments were used
Statistical Analysis 4: Comparison: Scar Negative Volume - Placebo vs Scar Negative Volume - 1 mg AZX100; Test type: Superiority or Other; p = 0.079, Wilcoxon (signed rank); For this early phase study, no adjustments were used
Statistical Analysis 5: Comparison: Scar Total Volume - Placebo vs Scar Total Volume - 0.3 mg AZX100; Test type: Superiority or Other; p = 0.16, Wilcoxon (signed rank); For this early phase study, no adjustments were used
Statistical Analysis 6: Comparison: Scar Total Volume - Placebo vs Scar Total Volume - 1 mg AZX100; Test type: Superiority or Other; p = 0.45, Wilcoxon (signed rank) — For this early phase study, no adjustments were used; For this early phase study, no adjustments were used

ADVERSE EVENTS:
Time Frame: Adverse events began to be collected for each patient after dosing with study agent, and were collected for the duration of the study (12 months). The adverse event collection period for the entire study lasted for a period of 15 months.
Arm/Group | Low Dose | High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 18/21 | 17/19 | 18/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=21) | High Dose (N=19) | Placebo (N=19)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (12) | 4 (4) | 4 (6)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 6 (10) | 8 (14) | 5 (9)
Injection Site Irritation (General disorders) | 8 (13) | 5 (11) | 5 (8)
Injection Site Pain (General disorders) | 6 (15) | 11 (19) | 8 (17)
Injection Site Pruritus (General disorders) | 4 (5) | 3 (4) | 4 (4)
Injection Site Reaction (General disorders) | 2 (2) | 0 (0) | 1 (1)
Injection Site Urticaria (General disorders) | 6 (11) | 9 (15) | 4 (5)
Nasopharyngitis (Infections and infestations) | 2 (4) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (6) | 2 (3) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less